CLINICAL TRIAL: NCT05628467
Title: Association Between Antidepressant Use and Falls in Older Adults: Analysis of the World Health Organization Global Database
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco20221004
Record Dates: First submitted 2022-10-27; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-10

CONDITIONS: Antidepressants Causing Adverse Effects in Therapeutic Use; Fall
MeSH Terms: interventions — Antidepressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antidepressive Agents — Compare the signal obtained from the pharmacovigilance database study between adults over 65 who fall on antidepressants versus those who fall on other drugs

SUMMARY:
The incidence of fall in older adults aged 65 and over is estimated at 30%, and 50% of the people aged 80 and over with at least one fall a year. Falls are associated with significant morbidity and mortality.

The origin falls is often multifactorial, involving intrinsic and extrinsic factors. Few studies have investigated the association with all antidepressants. Potential adverse effects of antidepressants such as hyponatremia, sedation, orthostatic hypotension, extrapyramidal symptoms are known risk factors for falls. Due to multimorbidity, polypharmacy including interaction risks, and aging-related changes in pharmacokinetic and pharmacodynamic of drugs, antidepressants may further increase this risk in older patients.

Based on the World Health Organization global database, the main objective of this study is to investigate the association between antidepressants classes and the occurrence of falls reported in the database.

A disproportionality analysis will be performed. It will aim to assess whether some classes of antidepressants, and within these classes some molecules, are associated with a greater risk of falls.

A mediation analysis will also be performed. It will aim to examine some of the mediators involved in the association between antidepressants classes and falls.

ELIGIBILITY:
Inclusion Criteria:

* be over 65 years old
* take antidepressants
* have already presented falls

Exclusion Criteria:

-

Ages: 65 Years to 120 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients aged 65 years and over who presented fall on antidepressants
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of the studied population | 01/07/2022
  The investigators describe the profile of patients who are reported in the WORLD HEALTH ORGANIZATION Vigibase pharmacovigilance database, as having experienced a fall. In particular, the number of patients who use antidepressants (Non-selective monoamine reuptake inhibitors, Selective serotonin reuptake inhibitors, Selective serotonin-norepinephrine reuptake inhibitors, Alpha-2-adrenergic receptor antagonists, Monoamine oxidase inhibitors, other antidepressants), the number of patients who presented associated illnesses known to induce falls, the number of patients who presented associated drug prescriptions known to induce falls.
Analysis of the association between antidepressant classes and falls reporting, among subjects aged 65 or older | 01/07/2022
  A disproportionality analysis is carried out in multivariate analysis, taking into account some confounding factors (potentially associated illnesses and prescriptions known to induce falls)

SECONDARY OUTCOMES:
Analysis by age group | 01/07/2022
  Investigators study the association between antidepressant classes and falls reporting for the age group 65-74 and for the age group 75 and over.
  A disproportionality analysis is carried out in multivariate analysis, taking into account some confounding factors (potentially associated illnesses and prescriptions known to induce falls)
Analysis of the most frequent antidepressants | 01/07/2022
  Investigators study the association between most frequent antidepressants and falls reporting among patients aged 65 or older.
  We identified most frequent antidepressants as those with more than 1000 cases reported in VigiBase®.
  A disproportionality analysis is carried out in multivariate analysis, taking into account some confounding factors (potentially associated illnesses and prescriptions known to induce falls)
Mediation analysis | 01/07/2022
  Investigators study the association between antidepressant classes and falls reporting analysing the potential role of hyponatraemia and delirium as mediators. This analysis is carried out taking into account some confounding factors (potentially associated illnesses and prescriptions known to induce falls)

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Department of Pharmacology, Caen, Normandy, France